CLINICAL TRIAL: NCT07173361
Title: Investigating the Impact of Micronized Progesterone on Skeletal Muscle Metabolism
Brief Title: Progesterone and Muscle Protein Synthesis in Premenopausal Women (MP4-MPS)
Acronym: MP4 MPS
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MP4-MPS
Record Dates: First submitted 2025-09-07; First posted 2025-09-15 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers; Female; Progesterone; Premenopausal
Keywords: Progesterone; Muscle protein synthesis; Stable isotope tracer; Female physiology; Premenopausal females; Exercise metabolism; Micronized progesterone; Resistance exercise; Skeletal muscle
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Intervention Model Description: Parallel assignment with within-participant leg comparison. Participants are randomized 1:1 to micronized progesterone or matched placebo and complete the same unilateral resistance exercise and infusion protocol. Both groups receive identical procedures; only the study drug differs. The exercised leg serves as an internal comparator to the contralateral rested leg for physiologic endpoints (this is not a crossover). Randomization is computer-generated with concealed allocation; study staff, participants, and outcome assessors are blinded to assignment. Single-site conduct.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Micronized Progesterone (Experimental): Drug - Micronized progesterone (oral capsules; 400 mg total as 2 × 200 mg at ~34 h and ~10 h pre-trial)
  Interventions: Drug: Micronized progesterone (oral capsules)
- Placebo Comparator: Placebo (Placebo Comparator): Drug - Placebo (oral capsules; matched schedule and appearance)
  Interventions: Drug: placebo capsule

INTERVENTIONS:
Drug: Micronized progesterone (oral capsules) — Two doses of 400 mg total micronized progesterone, administered as 2 × 200 mg capsules ~34 hours and ~10 hours prior to infusion trial, taken with a standardized nutritional drink.
  Other Names: PROMETRIUM
  Arms: Experimental: Micronized Progesterone
Drug: placebo capsule — Matched oral placebo capsules administered on the same schedule (~34 and ~10 hours prior to infusion trial) with a standardized nutritional drink.
  Arms: Placebo Comparator: Placebo

SUMMARY:
The goal of this clinical trial is to learn if micronized progesterone (PROMETRIUM®) influences the muscle-building response to resistance exercise in healthy premenopausal women aged 18-30 years.

The main questions it aims to answer are:

1. Does progesterone change the rate of muscle protein synthesis after exercise?
2. Does progesterone alter the difference in synthesis between an exercised leg and a rested leg?

Researchers will compare micronized progesterone to a placebo to see if progesterone changes the way skeletal muscle adapts to resistance exercise.

Participants will:

* Take two oral doses of progesterone (400 mg total, 34 and 10 hours before testing) or placebo
* Complete a unilateral leg extension exercise session in the lab
* Receive an infusion of a stable isotope tracer and provide blood samples
* Undergo muscle biopsies from the exercised and rested legs

DETAILED DESCRIPTION:
This is a single-site, randomized, double-blind, placebo-controlled Phase 1 clinical trial designed to evaluate the effects of micronized progesterone on exercise-induced skeletal muscle protein synthesis (MPS) in premenopausal women.

Participants will be healthy, naturally menstruating women aged 18-30 years. Each will be randomized to receive either two oral doses of micronized progesterone (400 mg total, administered as 2 × 200 mg capsules, 34 and 10 hours prior to testing) or a matched placebo.

During the infusion trial, participants will consume a standardized nutritional drink (~530 kcal; 22 g protein, 52 g carbohydrate, 26 g fat) and perform unilateral resistance exercise consisting of single-leg extensions (1 warm-up set followed by 4 working sets to volitional failure, 2-minute rest between sets).

To assess myofibrillar MPS, participants will undergo a primed continuous infusion of L-[ring-¹³C₆]-phenylalanine, with incorporation into muscle proteins determined from serial biopsies collected from both the exercised and rested legs. Blood samples will be obtained throughout the infusion period to measure plasma amino acids and hormone concentrations.

The primary endpoint is the treatment (placebo vs. progesterone) × leg (exercised vs. rested) interaction in MPS over the 5-hour post-exercise period. Secondary outcomes include the exercise-induced change in fractional synthetic rate (ΔFSR), plasma hormone responses, and exploratory measures of body composition and strength.

This study will provide direct evidence on whether progesterone modifies the acute anabolic response to resistance exercise in reproductive-age women, addressing an important gap in female skeletal muscle physiology.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identifies as female and is assigned female at birth.
2. Aged 18 to 30 years (inclusive).
3. Body mass index (BMI) between 18 and 34.9 kg/m² (inclusive).
4. In general, good health, as determined by a study-specific health screening questionnaire and medical history review.
5. Reports regular menstrual cycles (21-35 days in length) for the past 3 consecutive months.
6. Not currently using hormonal contraceptives and has completed a minimum 3-month washout period.
7. Resting blood pressure <140/90 mmHg at screening and on the infusion day.
8. Willing and able to provide written informed consent in English.

Exclusion Criteria:

1. Current use of tobacco, vaping products, or nicotine-containing substances.
2. Ineligible for physical activity as determined by the Get Active Questionnaire (GAQ).
3. Any medical, orthopedic, or psychiatric condition that, in the opinion of the Investigator, could interfere with the participant's ability to comply with study procedures or pose additional risk.
4. Current gastrointestinal or swallowing disorders that may interfere with supplement ingestion (e.g., chronic diarrhea, regurgitation, dysphagia).
5. Currently pregnant, planning to become pregnant, or known/suspected to be pregnant.
6. Use of hormonal contraceptives within the past 3 months.
7. Presence of any electronic medical devices or metallic implants that may interfere with DXA scanning or muscle biopsy procedures.
8. History of neuromuscular disorders or muscle/bone wasting diseases.
9. Current or recent use (within 3 months) of medications known to affect protein metabolism (e.g., glucocorticoids, systemic NSAIDs, isotretinoin, or anabolic agents).
10. Personal or first-degree family history of thrombotic events (e.g., DVT, PE, stroke, myocardial infarction).
11. Use of anticoagulant or antiplatelet medications.
12. Excessive alcohol intake (>21 units per week; 1 unit = 10 mL of pure ethanol).
13. History of bleeding disorders or known coagulation or platelet abnormalities.
14. Known hypersensitivity or allergy to micronized progesterone, soya, peanuts, or any excipients in the study capsule.
15. History or current diagnosis of liver dysfunction or hepatic disease, unless liver function tests have returned to normal ranges.
16. History or presence of contraindications to progesterone therapy, including any of the following:

    1. Known or suspected estrogen- or progestin-dependent malignancies (e.g., breast or endometrial cancer).
    2. History of endometrial hyperplasia or unexplained abnormal uterine bleeding.
    3. Active or prior history of arterial thromboembolic disease (e.g., stroke, myocardial infarction, coronary artery disease).
    4. History of classical migraine with aura.
    5. Active or prior history of venous thromboembolism (e.g., deep vein thrombosis, pulmonary embolism) or thrombophlebitis.
    6. History of partial or complete vision loss due to ophthalmic vascular events.
17. Clinically significant anemia or hematologic abnormalities (e.g., low hemoglobin or hematocrit) that may elevate the risk of biopsy complications.
18. Participation in another interventional study involving investigational drugs or invasive procedures within the past 30 days.
19. Documented history of severe vasovagal syncope or needle phobia that may interfere with study compliance or safety.
20. Known allergy or intolerance to any ingredient in the BOOST® 2.24 nutritional drink (e.g., milk protein, soy, corn-derived ingredients, cocoa, or artificial flavorings).

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Myofibrillar muscle protein synthesis (MPS) rate | 5 hours after standardized feeding and unilateral resistance exercise (infusion period)
  Incorporation of L-[ring-¹³C₆]-phenylalanine into myofibrillar proteins, measured via bilateral muscle biopsies (vastus lateralis, exercised vs. rested legs). The primary endpoint is the treatment (micronized progesterone vs. placebo) × leg (exercised vs. rested) interaction in MPS under fed conditions.

SECONDARY OUTCOMES:
Myofibrillar MPS in rested leg (fed condition) | 5 hours after standardized feeding
  MPS in the rested (non-exercised) leg to assess whether progesterone alters postprandial muscle anabolism in the absence of exercise.
Myofibrillar MPS in rested leg (fasted condition) | -240 to 0 minutes before feeding (fasted infusion period)
  MPS calculated from baseline fasted blood/plasma enrichment and pre-meal biopsy to determine whether progesterone alters basal, fasted-state anabolism.
Circulating serum progesterone concentrations (pharmacokinetics) | -240 to 300 minutes (fasted and fed infusion periods)
  Serial serum progesterone measured to characterize exposure; pharmacokinetic parameters include AUC, Cavg, Cmax, and Tmax.
Postprandial amino acid response | 0 to 300 minutes after standardized feeding
  Serial serum amino acid concentrations (including essential and branched-chain amino acids) measured for PK parameters (AUC, Cavg, Cmax, Tmax) to contextualize MPS responses.
Plasma tracer enrichment verification | Throughout infusion (-240 to 300 minutes)
  Plasma enrichment of L-[ring-¹³C₆]-phenylalanine at steady-state timepoints to confirm validity of MPS calculations (target ≥2.0%).
Baseline menstrual phase and hormonal status | Pre-dose (-240 minutes)
  Baseline serum estradiol, LH, and FSH concentrations to verify early follicular phase timing and ensure group comparability.

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Metabolism Research Laboratory, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the small sample size, the invasive nature of muscle biopsy procedures, and the risk of re-identification. Results will be disseminated in aggregate form through peer-reviewed publications and scientific presentations.